CLINICAL TRIAL: NCT06582277
Title: Phase 2a, Single Center, Randomized, Double-blind, Study to Evaluate the Immunogenicity and Safety of One Single Administration of OVX836 Influenza Vaccine at Two Dose Levels (180µg or 480μg) Given Intramuscularly (IM), Either as a Booster or a Primary Vaccination in Healthy Adults Previously Administered With OVX836, Influvac Tetra® or Placebo in the OVX836-002 (EudraCT Number: 2019-002939-28) and OVX836-003 (EudraCT Number: 2021-002535-39) Studies.
Brief Title: Safety and Immunogenicity of Two Dose Levels of OVX836 Influenza Vaccine as a Booster on Participants Previously Administered With OVX836
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Osivax (Industry)
Collaborators: Harmony Clinical Research BVBA (Other); Clinfidence (Unknown); Inferential (Industry); University Hospital, Ghent (Other); KCAS Bio (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: OVX836-007
Record Dates: First submitted 2024-08-26; First posted 2024-09-03 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Vaccine-Preventable Diseases; Influenza
MeSH Terms: conditions — Vaccine-Preventable Diseases; Influenza, Human

STUDY DESIGN:
Intervention Model Description: Randomized assignement to 2 dose-level of experimental vaccine (180µg and 480µg) in a 1:1 ratio for the booster group and open label assignement to 480µg dose of the experimental vaccine for the control group.
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- OVX836 - 180μg dose level (Experimental): 180 µg dose of an adjuvant-free recombinant influenza candidate vaccine based on the Nucleoprotein (NP) of the influenza virus.
  Interventions: Biological: OVX836 shot
- OVX836 - 480μg dose level (Experimental): 480 µg dose of an adjuvant-free recombinant influenza candidate vaccine based on the Nucleoprotein (NP) of the influenza virus.
  Interventions: Biological: OVX836 shot

INTERVENTIONS:
Biological: OVX836 shot — One single administration intramuscularly at Day 1.

SUMMARY:
This phase 2a is designed to evaluate the anamnestic response of a booster dose (either 180 µg or 480 µg) of OVX836 influenza vaccine administered intramuscularly to participants vaccinated three to five years ago in OVX836-002 or OVX836-003 studies. Participants who had received a placebo or Influvac Tetra® in previous studies would serve as controls and would receive the highest dose of OVX836 vaccine (480 µg) as a primary vaccination.

DETAILED DESCRIPTION:
This is a phase 2a, single center, randomized, double-blind study designed to evaluate the immunogenicity and safety of one single administration of OVX836 influenza vaccine at two dose levels (180μg or 480μg) given intramuscularly, either as a booster or a primary vaccination in approximately 160 to 220 healthy participants (aged 20-64 years) previously administered with OVX836, Influvac Tetra® or placebo in the OVX836-002 (EudraCT number: 2019-002939-28) and OVX836-003 (EudraCT number: 2021-002535-39) studies. This includes OVX836-002 participants who had received 180μg OVX836 during the influenza season 2019-2020 and OVX836-003 participants who had received 180μg, 300μg or 480μg OVX836 before the influenza season 2021-2022. Volunteers who received either Influvac Tetra® in the OVX836-002 study or a placebo in the OVX836-003 study will serve as controls and will receive a primary single dose of OVX836 480μg.

ELIGIBILITY:
Inclusion Criteria:

1. Subject who voluntarily provides written informed consent to participate in the study.
2. Healthy male or female subjects, as determined by medical history and medical examination
3. Subject compliant with the reproductive criteria for female participants
4. Subjects who participated in the OVX836-002 or OVX836-003 studies.
5. Subjects aged 20 and 64 years, inclusive.
6. Reliable and willing to commit to participating for the duration of the study, and capable of following study procedures diligently.
7. Ability and technical capability to complete an eDiary.

Exclusion Criteria:

1. Subjects with a body mass index (BMI) ≤18 kg/m² or ≥35 kg/m² on the day of vaccination.
2. Previous influenza vaccination within 6 months before the day of vaccination or planned to receive during the whole study period.
3. vaccination with an mRNA-based influenza vaccine including NP in its composition.
4. Any known or suspected immunodeficient conditions.
5. Past or current history of significant autoimmune diseases, as judged by the Investigator.
6. Current history of uncontrolled medical illness such as diabetes, hypertension, heart, renal or hepatic diseases.
7. Known or suspected infection with human immunodeficiency virus (HIV), hepatitis C virus (HCV), or hepatitis B virus (HBV).
8. Pregnant or lactating woman.
9. Female planning to become pregnant or planning to discontinue contraceptive precautions until the end of the trial.
10. Participants with extensive tattoos covering deltoid regions on both arms that would preclude the assessment of local reactogenicity.
11. Other vaccination within 3 months prior to the day of study vaccination for live attenuated vaccines, or within 1 month prior to the day of study vaccination for non-live vaccines, at the exception of COVID vaccines which can be administered within 14 days before or after study vaccine administration.
12. Planning to receive other vaccines during the first 28 days following the study vaccine administration.
13. Administration of any investigational or non-registered drug or vaccine within 3 months prior to the administration of study vaccines, or planned administration of any such product during the entire study period.
14. History of receiving blood, blood components or immunoglobulins within 3 months prior to the day of vaccination or planned to receive such product during the whole study period.
15. Presence of an acute febrile illness on the day of vaccination (oral temperature >38.0°C, temporary exclusion criterion).
16. Past or current history of any progressive or severe neurological disorder, seizure disorder or Guillain-Barré syndrome.
17. Behavioral or cognitive impairment, or psychiatric disease that, in the opinion of the Investigator, may interfere with the subject's ability to participate in the study.
18. History of alcohol or drug abuse that ceased less than 6 months before enrolment, current alcohol or drug abuse according to the Investigator's judgement), smoking habit of more than 10 cigarettes/day, or current vaping (nicotine consumption corresponding to more than 10 cigarettes/day).
19. Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs during the period starting 3 months before the study vaccine administration. For corticosteroids, this will mean prednisone equivalent ≥20 mg/day. Inhaled, topical and intra-articular steroids are allowed.
20. Current or past malignancy, unless completely resolved for >5 years (except non-metastatic basal cell carcinoma which has been completely resected).
21. History of severe allergic reactions and/or anaphylaxis, or serious adverse reactions to vaccines or allergy to kanamycin or any other component of the vaccine.
22. Any contraindication to IM administration, as judged by the Investigator.
23. Individuals with a history of any illness that, in the opinion of the Investigator, could potentially interfere with the results of the study or pose additional risk to the subjects by participating in the study.
24. Sponsor employees or Investigator site personnel directly affiliated with this study and their immediate families. Immediate family is defined as a spouse, parent, child or sibling, whether biological or legally adopted, including children of newly composed families.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 117 (Actual)
Dates: Start 2024-10-22 (Actual); Primary Completion 2025-06-02 (Actual); Study Completion 2025-06-02 (Actual)

PRIMARY OUTCOMES:
Safety evaluation of OVX836 (180µg and 480µg) | From enrollment to the end of trial at 180 days.
  Description: Proportion of subjects reporting: - solicited local and systemic symptoms within 7 days after vaccine administration - unsolicited AEs within 29 days after vaccine administration - SAEs during the entire study duration - ILIs and RT-PCR confirmed influenza A or B (overall and occurring more than 14 days post-vaccination, i.e., vaccine failure), RSV and/or SARS-CoV-2.

SECONDARY OUTCOMES:
Cell-mediated immune response to OVX836 (180μg and 480μg) in term of NPspecific IFNγ spot forming cells frequencies in peripheral blood (ELISPOT) | at Days 1, 8 and 29
Frequencies of NP-specific CD4+ and CD8+T-cells expressing IL-2, TNFα and/or IFNγ, measured by flow cytometry, following in vitro stimulation of PBMC | at Days 1, 8 and 29
Cross-reactivity of the NP influenza-specific responses by IFNγ ELISPOT against selected circulating and emerging strains of influenza | at Days 1, 8 and 29
Geometric mean titers (GMTs) of anti-NP Immunoglobulin G (IgG) (ELISA, serum) | at Days 1, 8 and 29
Number and percentage of subjects with an increase (two-fold and four-fold) in anti-NP IgG (ELISA, serum) | at Days 1, 8 and 29
GMTs of anti-OVX313 tag (Oligodom®) IgG level (ELISA, serum) | at Days 1, 8 and 29
Anti-C4bp (C4b-binding protein) oligomerization domain IgG titers (ELISA, serum) in subjects with positive result for anti-OVX313 (anti-OVX313 titer >12.5). | at Days 1, 8 and 29

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Groth, MD, Study Director — Osivax
Locations (1):
- Centre for Vaccinology (CEVAC) Ghent University Hospital, Ghent, Belgium

IPD SHARING:
Plan to Share IPD: No